CLINICAL TRIAL: NCT01892683
Title: Breath Monitoring of Propofol in Patients Undergoing Anesthesia for Surgical Procedures(Observational Study)
Brief Title: Breath Monitoring of Propofol (Observational Study)
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Cyrill Hornuss, Dr. Cyrill Hornuss, Ludwig-Maximilians - University of Munich
Other Study IDs: ExhaledPropofolPK
Record Dates: First submitted 2013-06-26; First posted 2013-07-04 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Anesthesia
Keywords: propofol; exhaled; monitoring; anesthesia
MeSH Terms: interventions — Anesthesia, General; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Propofol: This study will investigate patients that undergo routine anesthesia for elective surgical procedure at the hospital of the University of Munich(Klinikum der Universität München. Patients will receive intravenous anesthesia with propofol.
  Interventions: Drug: General anesthesia with propofol

INTERVENTIONS:
Drug: General anesthesia with propofol — Study subjects will undergo general anesthesia with propofol according to the clinical standard protocol practiced at the hospital of the University of Munich.
  Other Names: propofol-lipuro

SUMMARY:
This trial investigates the relationship between concentrations of the anesthetic drug propofol in exhaled breath and blood in patients undergoing general anesthesia for elective surgery. The main goal of this study is to develop a population pharmacokinetic model for propofol in exhaled breath.

DETAILED DESCRIPTION:
Propofol is a hypnotic drug commonly used for induction and maintenance of general anesthesia. Propofol is adiministered intravenously and has a comfortable side effect profile. Patients recover fast after propofol anesthesia and are less likely to suffer from post-operative nausea and vomiting compared to general anesthesia with inhalational anesthetics. However, titration of propofol can be challenging and patients may suffer from over- or underdosing during propofol anesthesia. Recent work has demonstrated that propofol is exhaled during anesthesia. Monitoring of propofol concentrations in breath gas during anesthesia may help to titrate propofol anesthesia more effectively. Yet, it is unclear how propofol concentrations vary among patients. This study aims to investigate this variation in a cohort of patients undergoing general anesthesia for elective surgical procedures. Propofol will be measured in breath gas continuously from the induction of anesthesia until recovery. Blood samples will be drawn from the start of anesthesia up to 24 h after the end of the anesthesia procedure and assayed for propofol blood concentrations. We will built a pharmacokinetic model from breath and blood measurements in order to describe the variability of propofol breath concentrations among study participants.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for routine surgery
* age ≥ 18 years
* planned duration of intervention > 1 hour
* written informed consent

Exclusion Criteria:

* propofol administration within 3 days prior to planned intervention
* pregnancy
* inability to give informed consent
* retraction of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study persons undergo general anesthesia for elective routine surgery at the hospital of the University of Munich (Klinikum der Universität München)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Exhaled Propofol | Continuous measurement during anesthetic procedure
  Propofol concentrations in breath gas will be assessed every 500 ms during the anesthesia procedure. Participants will be followed for the duration of the anesthesia procedure, an expected average of 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Cyrill Hornuss, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Klinikum der Universität München, Campus Großhadern, München, Bavaria, Germany

REFERENCES:
- [Background] Hornuss C, Praun S, Villinger J, Dornauer A, Moehnle P, Dolch M, Weninger E, Chouker A, Feil C, Briegel J, Thiel M, Schelling G. Real-time monitoring of propofol in expired air in humans undergoing total intravenous anesthesia. Anesthesiology. 2007 Apr;106(4):665-74. doi: 10.1097/01.anes.0000264746.01393.e0. PMID 17413903
- [Background] Hornuss C, Wiepcke D, Praun S, Dolch ME, Apfel CC, Schelling G. Time course of expiratory propofol after bolus injection as measured by ion molecule reaction mass spectrometry. Anal Bioanal Chem. 2012 Apr;403(2):555-61. doi: 10.1007/s00216-012-5856-3. Epub 2012 Feb 28. PMID 22370587